CLINICAL TRIAL: NCT02218892
Title: Prediction of Temporomandibular Involvement in Juvenile Idiopathic Arthritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Malin Collin (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Malin Collin, DDS, PhD-student, Folktandvården Stockholms län AB
Organization: Folktandvården Stockholms län AB (Other Government)
Other Study IDs: 2010/2089-31/2
Record Dates: First submitted 2014-06-30; First posted 2014-08-18 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Juvenile Idiopathic Arthritis; Temporomandibular Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum,saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Juvenil Idiopathic Arthritis: The group consists of children age 7-14 with an diagnosis of active Juvenile Idiopathic Arthritis.

SUMMARY:
Purpose and aims The general aim of this project is to improve the diagnostic methods for disease activity and identify predictive factors (clinical and radiographic factors, pro- and anti-inflammatory mediators in saliva and plasma) for temporomandibular joint (TMJ) involvement in juvenile idiopathic arthritis (JIA).

The hypothesis is that self-reported pain and impaired jaw function together with clinical findings correlates well with radiological signs of jaw involvement.

Null hypothesis: Self-reported pain, impaired jaw function and clinical findings do not correlate with radiological signs of jaw involvement.

Study 1 The aim of this study is to investigate which findings from the patient history and from clinical examination that is of significance for diagnostics of TMJ involvement in patients with JIA both in a short- and long-term perspective. The patients will be followed-up during two years. They will undergo a clinical examination according to Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD; Dworkin and LeResche 1992) once a year and a telephone follow-up sixth months after the clinical examination. Further, the clinical findings from the orofacial regions will be compared to their general disease activity.

Study 2 The aim of the second study is to correlate radiological findings and clinical findings in order to investigate any early radiological signs of disease activity and progression but also to compare the radiographic examination using conventional panoramic technique with computer tomography (CT).

DETAILED DESCRIPTION:
One-hundred consecutive patients with active JIA, as diagnosed by the Department of Pediatric Rheumatology, Astrid Lindgrens Barnsjukhus, Karolinska University Hospital will be included.

Inclusion criteria are:

* age between 7 and 14 years
* a diagnosis of JIA according to the International League of Associations for rheumatology

Exclusion criteria are:

* current malignancies
* TMJ surgery or trauma within two years
* recent intra-articular glucocorticoid injection in TMJ (within 1 month)
* other conditions or diseases than JIA that may cause orofacial pain. The parents of the patients and/or the patients will give their verbal and written informed consent to participate in the study according to the permission from the regional ethical committee 2011/2:1.

Clinical examination and follow-ups The patients will be examined clinically three times with an interval of 12 months. The clinical examination will be performed according to the RDC-TMD by calibrated investigators. Panoramic x-ray and CT scans will be performed at the inclusion examination as well as at the end of the study after 24 months. Pharmacological treatment will be recorded at every clinical examination and at telephone interviews. The patients will also be examined by a pediatric rheumatologist regarding general disease activity according to the Juvenile Arthritis Disease Activity Score 27 (JADAS-27), the Short Form (36) Health Survey (SF-36), thrombocyte particle count, C-reactive protein and blood titer of rheumatoid factor and anti-cyclic citrullinated peptides. Information from the examination by the pediatric rheumatologist will be drawn from the Swedish national register for children with JIA.

Telephone interview Six months after the first and second visit, a structured telephone interview with the patients and/or their parents will be performed according to a questionnaire. The objective is to estimate the degree of joint pain and functional limitations in jaw function.

Radiological examination Conventional panoramic x-rays and bilateral TMJ images will be obtained with the digital volume tomography (DVT, New Tom Model QR-DVT 9000, New Tom AG, Marburg, Germany). The CT sections will be evaluated by a specialist in oral radiology for presence of radiographic signs of cortical and subcortical erosions, flattening, sclerosis and ramus height.

ELIGIBILITY:
Inclusion Criteria:

1. age between 7 and 14 years
2. a diagnosis of JIA according to the International League of Associations for rheumatology (ILAR) The parents of the patients and/or the patients will give their verbal and written informed consent to participate in the study according to the permission from the regional ethical committee 2011/2:1.

Exclusion Criteria:

1. current malignancies
2. TMJ surgery or trauma within two years
3. recent intra-articular glucocorticoid injection in TMJ (within 1 month)
4. other conditions or diseases than JIA that may cause orofacial pain.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: One-hundred consecutive patients with active JIA, as diagnosed by the Department of Pediatric Rheumatology, Astrid Lindgrens Barnsjukhus, Karolinska University Hospital will be included.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2011-02; Primary Completion 2017-08 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Clinical findings in children with JIA | 2 years
  To find similarities in patients with JIA according to RDC-TMD (a clinical protocol validated for children)
Radiographic findings in children with JIA | Two years
  Repeated radiographic examination
Patient history | Two years
  Repeated interview on function and pain in the jaw area

CONTACTS AND LOCATIONS:
Overall Officials: Britt Hedenberg Magnusson, PhD DDS, Study Director — Karolinska Institutet
Locations (1):
- Folktandvården Stockholmslän AB, Stockholm, Sweden